CLINICAL TRIAL: NCT01629238
Title: Characteristics of Plant Sterols Consumers in France
Status: Completed | Type: Observational
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Other Study IDs: NU333
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular risk; dairy enriched product with plant sterols; general practitioners; adults followed by general practitioners
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group 1: group 1 = consumers of marketed drinkable low fat fermented milk enriched with plant sterol
- group 2: group 2 = non-consumers of marketed drinkable low fat fermented milk enriched with plant sterol

SUMMARY:
The purpose of this study is to describe the cardiovascular risk profile in subjects who consume a marketed drinkable low fat fermented milk enriched with plant sterol. Investigations are lead prospectively and retrospectively among adults enrolled from general practitioners' database.

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 18-70 years, regular visits to GP (at least once every six months within the past 2 years), agreeing to a written informed consent

Exclusion Criteria:

* any clinical, psychological or language problem that would prevent from completing the questionaires or communicating with GP

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults followed by general practitionners
Sampling Method: Non-Probability Sample
Enrollment: 780 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BKL Consultant, Boulogne-Billancourt, France